CLINICAL TRIAL: NCT03049345
Title: Gastric Cancer Sentinel Lymph Node Sampling: Refining Patient Selection for Organ Sparing Resection of Early Gastric Cancer in a North American Context
Brief Title: Gastric Cancer Sentinel Lymph Node Mapping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Carmen Mueller, Assistant Professor of Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-288-GEN
Record Dates: First submitted 2017-02-06; First posted 2017-02-10 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer; Sentinel Lymph Node; Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Radioactive Tracers; Methylene Blue

STUDY DESIGN:
Intervention Model Description: human subjects
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel Node Sampling Arm (Experimental): The day before surgery, 2mL of endoscopically-placed technetium 99m sulfur colloid solution will be injected submucosally at 4 points around the tumour. At the time of surgery, 2cc of 1% isosulfan blue dye will be similarly injected. Laparoscopically, the gastrocolic ligament will be opened to expose all gastric lymph node drainage basins. Using visual inspection and a laparoscopic gamma probe, blue nodes and those emitting 10x greater than background activity will be considered sentinel nodes and extracted. Patients will then under regular gastric cancer resection with D2 lymphadenectomy as per routine in our institution.
  Interventions: Procedure: Sentinel Lymph Node Sampling; Drug: Radioactive Tracers; Drug: Methylene Blue 20 MG/ML

INTERVENTIONS:
Procedure: Sentinel Lymph Node Sampling — The day before surgery, 2mL of endoscopically-placed technetium 99m sulfur colloid solution will be injected submucosally at 4 points around the tumour. At the time of surgery, 2cc of 1% isosulfan blue dye will be similarly injected. Laparoscopically, the gastrocolic ligament will be opened to expose all gastric lymph node drainage basins. Using visual inspection and a laparoscopic gamma probe, blue nodes and those emitting 10x greater than background activity will be considered sentinel nodes and extracted. Sentinel lymph nodes and resected specimens will be analyzed by permanent section.
Drug: Radioactive Tracers — see above
Drug: Methylene Blue 20 MG/ML — see above

SUMMARY:
Gastric cancer has an incidence in North America of over 24,000 new cases annually, of which approximately 15% are diagnosed at an early stage. Standard of care for early gastric cancer (EGC) treatment has historically included anatomical resection with regional lymphadenectomy. However, with the recent emergence of organ-sparing techniques, select patients with a very low risk of lymph node metastases are able to avoid anatomical resection and its inherent short and long term consequences. Despite this advance, EGC patients with high risk features continue to require anatomical resection to achieve adequate lymph node staging, despite the fact that 75-95% of these patients ultimately are found to have node negative disease. Due to the inadequacy of standard imaging modalities to reliably detect nodal metastases in EGC patients, sentinel lymph node sampling for gastric cancer was developed using principals similar to those used broadly for breast and melanoma patients. Early reports from Asia suggest this technique has very high success rates, accuracy and sensitivity, however it has never been verified in a North American context. This study aims to test SLN sampling for North American gastric cancer patients at a high volume regional treatment centre, with an aim to expand the application of organ sparing resection to EGC patients.

This project aims to determine the sensitivity and accuracy of sentinel lymph node sampling for early gastric cancer patients at a high volume, North American, tertiary care centre.

DETAILED DESCRIPTION:
Gastric cancer incidence in North America is 7.4/100,000 population, with 24,590 new cases diagnosed annually in the United States1. Of these, approximately 15% are detected at the early gastric cancer stage with no spread to regional lymph nodes2. Recent advances in gastric cancer detection, such as endoscopic use of narrow band imaging and magnification endoscopy, can help improve the detection rate of early lesions3-5. Gastric cancers detected at an early stage have an excellent prognosis, with reported long term overall survival rates of 71-92%6-9 due to the low rate of peritoneal and distant metastatic spread which frequently occur in patients with more advanced lesions. However, the mainstay of treatment even for early gastric cancers (EGC) remains anatomical resection with regional lymphadenectomy. While oncologically sound, anatomical resection is often associated with complications and unpleasant short and long-term side effects, including post-operative weight loss, dumping syndrome, vitamin deficiencies, anastomotic complications, delayed gastric emptying, and bile reflux, among others. Given the long life expectancy of patients after resection of EGC, curative resection with organ preservation to improve post-operative quality of life should be a treatment goal.

Recently, organ-sparing techniques have emerged which allow select early gastric cancers to be treated without anatomical resection. These techniques, including endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD), allow for curative resection of highly-selected lesions with complete organ preservation. The shortcoming of all organ sparing resection techniques presently is that lymphadenectomy is not performed, leading some patients to perhaps be under-staged and therefore under-treated.

According to the Japanese Gastric Cancer Treatment Guidelines10, early lesions are deemed appropriate for organ-sparing endoscopic resection if they meet the following criteria: confined to the mucosa (T1a), tumour size <2cm, no ulceration, and well-differentiated tumour grade. Together, tumours with these features have a very low risk of lymph node metastases (<1%). Long-term outcomes of ESD are highly favorable, with local recurrence and overall survival rates comparable to anatomical resection7,8. For tumours that do not meet the above criteria however, risk of lymph node involvement is drastically increased, with submucosal invasion, ulceration, tumour size >3cm, poorly differentiated tumour type, and lymphovascular invasion conferring a risk of lymphatic metastases of 4-26%11. For this reason, current best practices recommend EGCs with high risk features continue to undergo anatomical resection with regional lymphadenectomy. However 75-95% of such patients will ultimately have no regional metastases on final pathological analysis, suggesting they could have been spared anatomical resection if only their lymph node basins had been definitively staged prior to surgery.

Presently, several imaging modalities are available to characterize lymph node stage for gastric cancer, including endoscopic ultrasound (EUS), computed tomography (CT) and positron emission tomography (PET). Unfortunately, the sensitivity of these modalities is woefully inadequate to accurately predict microscopic lymph node metastases, and therefore they cannot be reliably used to differentiate high risk EGCs that require anatomical resection and lymphadenectomy from those amenable to organ-sparing resection12-15.

To address this gap in the ability to accurately detect nodal metastases in early gastric cancer, sentinel lymph node (SNL) sampling was pioneered in Asia and has undergone refinement and study there since the early 2000s. A recent multi-institutional study of 397 patients conducted across 12 centres in Japan reported rates of SLN detection of 97.5% and accuracy of SLN stage when compared to post-resection stage of 99%16. These numbers rival those reported for SLN biopsy of breast and melanoma cancers in large randomized controlled trials17,18. Indeed, for these tumour types, SLN biopsy is now the standard of care globally for staging clinically node-negative patients due to its diagnostic superiority over other staging modalities. Following the success of SLN sampling in gastric cancer, select Asian institutions are now applying this technique to diverting sentinel node-negative (SLN -ve) T1 and T2 gastric cancer patients away from anatomical resection with extensive lymphadenectomy and towards organ-sparing endoscopic or wedge resection.

The Upper GI Oncology Program at the McGill University Health Centre sees approximately 80 gastric cancer patients per year, in whom SLN sampling has the potential to inform resection decisions ~25-30%. Currently, the program performs 15-20 ESDs annually for both early esophageal and gastric lesions, and approximately 30-40 anatomical resections are performed in node-negative gastric and esophageal cancer patients per year. Implementation of the gastric SNL sampling technique would enable expansion of the ESD program to offer organ-sparing curative resections to EGC patients who presently can only be offered anatomical resection.

The purpose of this study is to determine the utility and feasibility of SLN sampling for gastric cancer in a North American context.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are deemed healthy enough to withstand laparoscopic or open anatomic gastrectomy with extended regional (D2) lymphadenectomy will be eligible. Patients much have biopsy-proven, single lesion, <4cm gastric adenocarcinoma, of stage cT1/T2/T3 N0 M0.

Exclusion Criteria:

* Not able to withstand anatomical gastric resection with D2 lymphadenectomy, patient refusal, N+ve disease on pre-op work up, disease progression before surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients in whom sentinel lymph node status accurately predicts true nodal status after anatomical gastrectomy and complete pathological examination | 3-4 weeks after study completion
  The % of patients in whom SLN status matched nodal status overall will be calculated
Sensitivity of Sentinel Lymph Node Sampling Method | 3-4 weeks after study completion
  # of patients with +ve SLN / # of patients with +ve lymph nodes in total
Specificity of Sentinel Lymph Node Sampling Method | 3-4 weeks after study completion
  # of patients with -ve SLNs / # of patients with -ve lymph nodes in total

SECONDARY OUTCOMES:
Adverse events due to SLN sampling technique | at time of surgery
  Complications of SLN intervention (allergic reaction, intra-operative bleeding, conversion to open approach)
Length of stay | 90 days from study completion
  # of days patient stays in hospital after procedure
R0 Resection rate | 3-4 weeks after study completion
  # of patients who have complete measurable disease excision at time of surgery
3 year Disease free survival rate | 3 years after study completion
  # of patients who are free of gastric cancer at 3 years out of all study patients
conversion to open | at time of surgery
  Number of patients who required a conversion to open technique after starting laparoscopically
Patient mortality | 90 days after surgery
  # of patients who die within 30 days of surgery or who die while in hospital
3 year overall survival rate | 3 years after study completion
  number of patients who are still alive at 3 years out of all study patients
Adverse surgical events | 30 days after study completion
  # of patients who suffered any of the following surgical complications: urinary tract infection, pneumonia, ileus, anastomotic leak, reoperation within 30 days of surgery, readmission within 30 days of discharge, myocardial infarction, venous thromboembolism, bleeding requiring blood transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitagawa Y, Takeuchi H, Takagi Y, Natsugoe S, Terashima M, Murakami N, Fujimura T, Tsujimoto H, Hayashi H, Yoshimizu N, Takagane A, Mohri Y, Nabeshima K, Uenosono Y, Kinami S, Sakamoto J, Morita S, Aikou T, Miwa K, Kitajima M. Sentinel node mapping for gastric cancer: a prospective multicenter trial in Japan. J Clin Oncol. 2013 Oct 10;31(29):3704-10. doi: 10.1200/JCO.2013.50.3789. Epub 2013 Sep 9. PMID 24019550
- [Background] Gotoda T, Yanagisawa A, Sasako M, Ono H, Nakanishi Y, Shimoda T, Kato Y. Incidence of lymph node metastasis from early gastric cancer: estimation with a large number of cases at two large centers. Gastric Cancer. 2000 Dec;3(4):219-225. doi: 10.1007/pl00011720. PMID 11984739
- [Derived] Mueller CL, Lisbona R, Sorial R, Siblini A, Ferri LE. Sentinel Lymph Node Sampling for Early Gastric Cancer-Preliminary Results of A North American Prospective Study. J Gastrointest Surg. 2019 Jun;23(6):1113-1121. doi: 10.1007/s11605-018-04098-5. Epub 2019 Mar 11. PMID 30859424